CLINICAL TRIAL: NCT06632769
Title: Continuous Monitoring of Body Temperature in Neonates During Skin-to-skin Care Immediately After Cesarean Section (MonT Neo) - a Prospective Observational Pilot Study
Brief Title: Continuous Monitoring of Body Temperature in Neonates During Skin-to-skin Care Immediately After Cesarean Section (MonT Neo)
Acronym: MonT Neo
Status: Completed | Type: Observational
Sponsor: Medical University of Graz (Other)
Responsible Party: Sponsor
Other Study IDs: MonTNeo
Record Dates: First submitted 2024-10-07; First posted 2024-10-09 (Actual); Last update posted 2025-07-10 (Actual); Status verified 2025-07

CONDITIONS: Body Temperature Measurement
Keywords: monitoring; body temperature; term neonates; transition; skin-to-skin care; Cesarean section

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- term neonates: term neonates after Cesarean section
  Interventions: Device: No intervention

INTERVENTIONS:
Device: No intervention — No intervention

SUMMARY:
The objective of this prospective observational pilot study is to apply the adhesive thermometer SteadyTemp® (SteadySense GmbH, Graz, Austria) in term neonates to monitor their body temperature non-invasively and continuously during skin-to-skin care with their mothers after Cesarean section and to compare these data with the one-time manual measurement of rectal body temperature as gold standard.

DETAILED DESCRIPTION:
Primary aim: To apply the adhesive thermometer SteadyTemp® (SteadySense GmbH, Graz, Austria) in term neonates in the right axillary area immediately after birth and to monitor their body temperature continuously during skin-to-skin care with their mothers after Cesarean section for 15 minutes.

Secondary aim

* To compare the body temperature with manually measured rectal temperature (single measurement).
* To examine the skin condition under the adhesive patch after 15 minutes of application using the Neonatal Skin Condition Scale (NSCS)17.

ELIGIBILITY:
Inclusion Criteria:

* Term neonates after caesarean section receiving skin-to-skin care immediately after birth
* Parental written informed consent

Exclusion Criteria:

* Preterm birth
* Need for respiratory support after birth
* No decision to conduct full life support
* No written informed consent
* Congenital malformation

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: term neonates born per caesarean section immediately after birth
Sampling Method: Non-Probability Sample
Enrollment: 40 (Actual)
Dates: Start 2024-10-24 (Actual); Primary Completion 2025-04-28 (Actual); Study Completion 2025-04-28 (Actual)

PRIMARY OUTCOMES:
body temperature | up to 15 minutes after birth
  body temperature continuously measured with SteadyTemp® (SteadySense GmbH, Graz, Austria)

CONTACTS AND LOCATIONS:
Locations (1):
- Medical University Graz, Graz, Styria, Austria

IPD SHARING:
Plan to Share IPD: Undecided
We need Data transfer agreement, before we can share our study data